CLINICAL TRIAL: NCT00058734
Title: Immune Responses to Antigen-Bearing Dendritic Cells in HIV-Infected Individuals
Brief Title: Therapeutic Vaccination Followed by Treatment Interruption in HIV Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01AI044628 (NIH); R01AI044628 (NIH)
Record Dates: First submitted 2003-04-11; First posted 2003-04-14 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: Dendritic Cell; Immunotherapy; Acute HIV; Human Immunodeficiency Virus; AIDS; HIV Therapeutic Vaccine; Treatment Experienced; Treatment Interruption
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — HIV Antigens

INTERVENTIONS:
Biological: Dendritic Cells Pulsed with HIV antigens

SUMMARY:
The aim of this trial is to find out if immune responses to HIV can be boosted in individuals who start medicines soon after being infected. If immune responses can be boosted to the virus, this may allow the body to control HIV without the need for medications. This study is designed to test a new strategy for boosting immune responses to HIV and to evaluate if these responses allow people to have control of HIV without medicines.

DETAILED DESCRIPTION:
The novel strategy used in this trial is to mix a peptide vaccine with dendritic cells from individuals. The dendritic cells are normal cells in the blood that boost immune responses. In HIV uninfected people, dendritic cells have been found to strongly activate the types of immune responses that may be important in controlling HIV.

HIV infected and HIV uninfected individuals in this study will receive one shot of dendritic cells alone followed by three monthly shots of dendritic cells plus vaccine. We will monitor the immune responses to the peptide vaccine during this time period. After completing the vaccinations, HIV infected patients will stop their HIV medications and their immune status (CD4 count) and viral load will be monitored closely over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Both HIV infected and HIV uninfected individuals are eligible for this study.

* CD4 cell count of 400 cells/mm3 or greater at study entry
* If HIV infected, initiated anti-HIV medicines within 120 days of infection
* If HIV infected, HIV viral load < 50 copies/ml for at least 3 months prior to study entry
* Current medication regimen for at least 3 months prior to study entry
* A particular blood type (HLA-A*0201)
* Acceptable methods of contraception

Exclusion Criteria:

* Received investigational drug or vaccine within 30 days prior to study entry
* On other immune-based therapy (e.g., interleukin-2, alpha interferon, immunoglobulin, thalidomide) within 30 days prior to study entry
* Megesterol acetate within 30 days prior to study entry
* Immunization within 4 weeks of study entry
* If hepatitis B virus (HBV) uninfected and at high risk for HBV infection, the patient will not be eligible until he or she has completed an HBV vaccine series.
* Unstable or severe medical condition, including active opportunistic infection requiring treatment
* History of Hashimoto's thyroiditis
* Cancer requiring chemotherapy within 6 months prior to study entry
* History of radiation therapy to axillary lymph nodes
* Significant laboratory abnormalities at study entry
* Pregnant or breastfeeding
* History of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, autoimmune hepatitis, scleroderma, mixed connective tissue disorder)
* Allergy to gentamicin, tobramycin, streptomycin, or amikacin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — New York University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dhodapkar MV, Steinman RM, Sapp M, Desai H, Fossella C, Krasovsky J, Donahoe SM, Dunbar PR, Cerundolo V, Nixon DF, Bhardwaj N. Rapid generation of broad T-cell immunity in humans after a single injection of mature dendritic cells. J Clin Invest. 1999 Jul;104(2):173-80. doi: 10.1172/JCI6909. PMID 10411546
- [Background] Dhodapkar MV, Krasovsky J, Steinman RM, Bhardwaj N. Mature dendritic cells boost functionally superior CD8(+) T-cell in humans without foreign helper epitopes. J Clin Invest. 2000 Mar;105(6):R9-R14. doi: 10.1172/JCI9051. PMID 10727452
- [Background] Larsson M, Jin X, Ramratnam B, Ogg GS, Engelmayer J, Demoitie MA, McMichael AJ, Cox WI, Steinman RM, Nixon D, Bhardwaj N. A recombinant vaccinia virus based ELISPOT assay detects high frequencies of Pol-specific CD8 T cells in HIV-1-positive individuals. AIDS. 1999 May 7;13(7):767-77. doi: 10.1097/00002030-199905070-00005. PMID 10357375
- [Background] Rosenberg ES, Altfeld M, Poon SH, Phillips MN, Wilkes BM, Eldridge RL, Robbins GK, D'Aquila RT, Goulder PJ, Walker BD. Immune control of HIV-1 after early treatment of acute infection. Nature. 2000 Sep 28;407(6803):523-6. doi: 10.1038/35035103. PMID 11029005